CLINICAL TRIAL: NCT03672539
Title: A Pilot Study of Liposomal Cytarabine and Daunorubicin (CPX-351) in Combination With Gemtuzumab Ozogamicin (GO) in Relapsed Refractory Patients With Acute Myeloid Leukemia (AML) and Post-Hypomethylating Agent (Post-HMA) Failure High-Risk Myelodysplastic Syndrome (HR-MDS)
Brief Title: Liposome-encapsulated Daunorubicin-Cytarabine and Gemtuzumab Ozogamicin in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) or High Risk Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0235; NCI-2018-01812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0235 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Gemtuzumab; CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPX-351, gemtuzumab ozogamicin) (Experimental): INDUCTION CYCLE: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 of cycle 1 and days 1 and 3 of cycle 2 and gemtuzumab ozogamicin IV over 120 minutes on day 1. Treatment repeats every 28 days for up to 2 cycles in the absence of unacceptable toxicity.
  CONSOLIDATION CYCLE: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 and gemtuzumab ozogamicin over 120 minutes on day 1. Treatment repeats every 28 days for up to 2 cycles in the absence of unacceptable toxicity.
  MAINTENANCE CYCLE: Patients receive gemtuzumab ozogamicin IV over 120 minutes on day 1. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the side effects and how well liposome-encapsulated daunorubicin-cytarabine and gemtuzumab ozogamicin work in treating patients with acute myeloid leukemia that has come back (relapsed) or that does not respond to treatment (refractory) or high risk myelodysplastic syndrome. Drugs used in chemotherapy, such as liposome-encapsulated daunorubicin-cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to a toxic agent called calicheamicin. Gemtuzumab ozogamicin attached to CD33 positive cancer cells in a targeted way and delivers calicheamicin to kill them. Giving liposome-encapsulated daunorubicin-cytarabine and gemtuzumab ozogamicin together may be an effective treatment for relapsed or refractory acute myeloid leukemia or high risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of liposome-encapsulated daunorubicin-cytarabine (liposomal cytarabine and daunorubicin [CPX-351]) in combination with gemtuzumab ozogamicin (GO) in relapsed refractory (R-R) patients with acute myeloid leukemia (AML) and post-hypomethylating agent (post-HMA) failure high-risk myelodysplastic syndrome (HR-MDS).

II. To determine the efficacy of liposomal cytarabine and daunorubicin (CPX-351) in combination with gemtuzumab ozogamicin (GO) in relapsed refractory patients with acute myeloid leukemia (AML) and post-hypomethylating agent (post-HMA) failure high-risk myelodysplastic syndrome (HR-MDS).

SECONDARY OBJECTIVE:

I. To determine the preliminary assessment of efficacy by response to revised International Working Group (IWG) criteria and time to response variables including overall survival (OS), event-free survival (EFS) and duration of response (DOR) of patients treated with this combination.

EXPLORATORY OBJECTIVES:

I. To determine the minimal residual disease (MRD) after treatment with this combination and its impact in long-term outcome.

II. To determine the effect of the level of pre-treatment expression of CD33 with response to this combination.

III. To determine the baseline CD33 genotype via CD33 polymorphism study, and its effect on response to this combination.

IV. To determine the effect of this treatment combination on responding patients transitioning to hematopoietic stem cell transplantation (HSCT).

V. To evaluate the effect of the treatment combination on Health Related Quality of Life (HRQoL) parameters.

OUTLINE:

INDUCTION CYCLE: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 of cycle 1 and days 1 and 3 of cycle 2 and gemtuzumab ozogamicin IV over 120 minutes on day 1. Treatment repeats every 28 days for up to 2 cycles in the absence of unacceptable toxicity.

CONSOLIDATION CYCLE: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 and gemtuzumab ozogamicin over 120 minutes on day 1. Treatment repeats every 28 days for up to 2 cycles in the absence of unacceptable toxicity.

MAINTENANCE CYCLE: Patients receive gemtuzumab ozogamicin IV over 120 minutes on day 1. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD33 positive (>= 3%), relapsed refractory acute myeloid leukemia by World Health Organization (WHO) criteria. Patients with post-hypomethylating agent (post-HMA) failure high-risk myelodysplastic syndrome (MDS), as defined by the presence of > 10% blasts, are also eligible.
* Patients with MDS or chronic myelomonocytic leukemia (CMML) who received hypomethylating agent based-therapy for the MDS or CMML and progress to AML are eligible at the time of diagnosis of AML regardless of any prior therapy for MDS or CMML. The WHO classification will be used for AML.
* Eastern Cooperative Oncology Group (ECOG) performance status score of =< 2.
* Total serum bilirubin =< 2 x upper limit of normal (ULN). Patients with known Gilbert's syndrome may have a total bilirubin up to =< 3 x ULN.
* Serum creatinine =< 2.0 mg/dl.
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 3 x ULN; =< 5 x ULN in case of suspected leukemic liver involvement.
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (b-HCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug. Effective methods of birth control include: Birth control pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin); intrauterine devices (IUDs); condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide; abstinence.
* Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation, oophorectomy, and/or hysterectomy.
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug.
* Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

* History of another primary invasive malignancy that has not been definitively treated and in remission. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses).
* Presence of clinically significant uncontrolled central nervous system (CNS) pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
* Evidence of active cerebral/meningeal disease. Patients may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of consent with at least 2 consecutive spinal fluid negative assessments for residual leukemia and negative imaging (imaging required only if previously showing evidence of CNS leukemia not otherwise documented by spinal fluid assessment).
* Patients with active unstable angina, concomitant clinically significant active arrhythmias, myocardial infarction within 6 months, or congestive heart failure New York Heart Association class III-IV. Patients with a cardiac ejection fraction (as measured by either multigated acquisition scan [MUGA] or echocardiogram) < 50% are excluded.
* Patients with total cumulative doses of non-liposomal daunorubicin, or other anthracycline equivalent, greater than 200 mg/m^2.
* Patients with uncontrolled, active infections (viral, bacterial, or fungal).
* Known active hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV).
* Patients with liver cirrhosis or other serious active liver disease or with suspected active alcohol abuse.
* Allogeneic hematopoietic stem cell transplantation (HSCT) within 6 months before the start of protocol-specified therapy, or with active acute/chronic graft-versus-host disease (GvHD) requiring systemic treatment; or receiving immunosuppression for GvHD prophylaxis within 2 weeks from the start of study therapy.
* Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exception: To reduce the circulating blast count or palliation; single dose intravenous cytarabine or hydroxyurea. No washout necessary for these agents.
* Patients must have recovered from acute non hematologic toxicity (to =< grade 1) of all previous therapy prior to enrollment.
* Females who are pregnant or lactating.
* Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards.
* Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
* Prior treatment with CPX-351 or gemtuzumab ozogamicin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 56 days
  Will use the Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia and Myelodysplasia. Will estimate the ORR for the combination treatment, along with the 95% credible interval.
Incidence and severity of all adverse events assessed using Common Toxicity Criteria version 4.0 | Up to 14 months

SECONDARY OUTCOMES:
Demographic/clinical characteristics (i.e. duration of response) and safety data of the patients | Up to 14 months
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.
Response and patient's clinical characteristics | Up to 14 months
  Will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate (Responders vs Non-Responders). Toxicity type, severity and attribution will be summarized for each patient using frequency tables.
Event-free survival | Up to 14 months
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Overall survival | Up to 14 months
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yesid Alvarado-Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org